CLINICAL TRIAL: NCT00551395
Title: Timing of Treatment Completion in Staged Selective Laser Trabeculoplasty (SLT): Early vs. Late Completion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Robert Campbell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC-1
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma
Keywords: glaucoma; laser; trabeculoplasty
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLT Early Completion (Arm 1) (Experimental): Intervention: 180 degrees of laser on Day 1, 180 degrees of laser on the other 180 degree on Day 2
  Interventions: Procedure: selective laser trabeculoplasty - early completion
- SLT Late Completion (Arm 2) (Active Comparator): Intervention: 180 degrees of laser on Day 1, 180 degrees of laser on the other 180 degrees at 1 month follow up appointment.
  Interventions: Procedure: Selective laser trabeculoplasty - late completion

INTERVENTIONS:
Procedure: selective laser trabeculoplasty - early completion — 180 degrees of laser on day 1 and other 180 degrees on day 2.
  Arms: SLT Early Completion (Arm 1)
Procedure: Selective laser trabeculoplasty - late completion — 180 degrees of laser on day 1 and other 180 degrees at 1 month follow up point.
  Arms: SLT Late Completion (Arm 2)

SUMMARY:
This study will evaluate the effect of the timing of treatment completion in two-staged selective laser trabeculoplasty therapy on intraocular pressure lowering effect.

DETAILED DESCRIPTION:
SLT therapy is used as an IOP lowering agent in patients with glaucoma. It is unknown whether the timing of a 2-staged approach to the laser therapy will result in better IOP lowering effect.

This study will evaluate the timing (early vs. late completion of SLT therapy) and determined the IOP lowering effect following the interventions.

Arm 1: Early Completion SLT

180 degrees of SLT on Day 1, 180 degrees of SLT on the other 180 degrees on Day 2

Arm 2: Late Completion SLT

180 degrees of SLT on Day 1, 180 degrees of SLT on the other 180 degrees at the 1 month follow up visit.

Primary Outcome: IOP (mmHg).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* primary open angle glaucoma or pseudoexfoliation glaucoma

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
intraocular pressure lowering | 1 month following procedure

SECONDARY OUTCOMES:
intraocular pressure lowering | 3, 6, 12 and 24 months following procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Campbell, MD, Principal Investigator — Queen's University, Kingston, Canada
Locations (1):
- Hotel Dieu Hospital & Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114